CLINICAL TRIAL: NCT02192021
Title: Phase I, Single-Arm, Open-Label, Dose Escalation Trial of MNA-Doxorubicin (MNA-D) in Patients-Subjects With Cutaneous T-cell Lymphoma (CTCL)
Brief Title: Micro Needle Array-Doxorubicin (MNA-D) in Patients With Cutaneous T-cell Lymphoma (CTCL)
Acronym: MNA-D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Falo, Louis, MD (Other)
Responsible Party: Principal Investigator, Oleg E. Akilov, MD, PhD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19080323
Record Dates: First submitted 2014-07-10; First posted 2014-07-16 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cutaneous T Cell Lymphoma
Keywords: CTCL; Cutaneous T-cell Lymphoma; Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Transdermal Patch; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Micro needle array-Doxorubicin (MNA-D) (Experimental): MNA-D application for all subjects
  Interventions: Drug: Micro needle array-Doxorubicin (MNA-D)

INTERVENTIONS:
Drug: Micro needle array-Doxorubicin (MNA-D) — MNA-D patches will be applied to 3-4 CTCL skin patches or plaques at each weekly visit (4/cycle). The initial safety, dose-finding phase will include one cycle of applications and the second phase will include weekly applications (4/cycle) for up to 6-8 cycles.
  Other Names: patch; doxorubicin

SUMMARY:
The study hypothesis is that in situ MNA-directed chemo-immunotherapy using doxorubicin will kill tumor cells locally and alter the tumor microenvironment to induce durable systemic tumor-specific immunity.

The purpose of this study is to test a new method of experimental treatment for CTCL, using small adhesive-like patches (a micro-needle applicator or MNA for short), which have dozens of very small micro-needles loaded with extremely low doses of doxorubicin, a chemotherapy agent. The overall goal of this study is to test the safety and effectiveness of these patches. We also want to determine which micro-dose of the drug is the best to achieve the best response. To make sure that we observe the effects of the very low dose of the drug and not the MNA patch itself, we will also use a placebo (a patch without drug in some patients) in addition to the doxorubicin coated patches. We will thoroughly evaluate the skin where the patches are applied. Once the best dose is determined for use in the patch, we will also begin to look at how well the patches work in clearing the skin.

DETAILED DESCRIPTION:
This study will evaluate a novel approach to the treatment of patches and plaques in the skin of patients diagnosed with cutaneous t-cell lymphoma utilizing a dissolvable microneedle array (MNA) delivery device that is used to directly and specifically deliver a drug to the tumor microenvironment for skin cancer therapy. We will utilize MNAs to deliver a well-characterized, potent chemotherapeutic agent (doxorubicin) to kill topically accessible, cutaneous T-cell lymphoma cells. In addition to directly killing cancer cells, doxorubicin is known to induce an immunologic cell death with the potential to simultaneously convert a cutaneous neoplasm into a highly potent patient specific immunogen capable of inducing innate, adaptive, and tumor specific effector and memory immune responses. Importantly, doxorubicin is currently in clinical use with a well-established safety profile. It is anticipated that use of the MNA-Doxorubicin (MNA-D) delivery system will enable direct and specific delivery of chemotherapy to the tumor, thereby avoiding any potential for systemic toxicity. The study will be conducted in two phases, with the first being a safety dose-finding phase and the second phase for efficacy and safety evaluation. The first phase is now completed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cutaneous T-cell Lymphoma (CTCL) based upon a skin biopsy diagnostic of atypical epidermotropism of folliculocentric or epidermotropic T-cells.
* Current stage of IA or IB.
* Expected survival of greater than or equal to12 months.
* Not be on any other investigational device/drug treatment.
* Have a sufficient number (i.e., n=4 for first dose cohort in Initial Safety Evaluation; n=3 for remainder of subjects) and surface area (> 5 cm2) of CTCL patches or plaques for Micro needle array-Doxorubicin (MNA-D) and Micro needle array (MNA) application.
* Willing to adhere to the instructions of the Investigator and his research team and sign an Informed Consent Form prior to entry into the study.
* Have the following initial and subsequent pretreatment laboratory parameters: granulocytes ≥2,000/mm3; platelets >50,000/mm3; serum creatinine ≤2X the upper limit of normal (ULN); AST, ALT, , LDH, Alk phos ≤3X the ULN.Subjects must be ³ 18 years of age and must be able to understand the written informed consent/assent document.
* Have no evidence of active infection, regardless of the degree of severity or localization. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible for study participation after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics before beginning treatment.
* Not receive any other treatment for CTCL except emollients of subject's choice without topical steroids, anti-fungal or antibacterial topical preparations.
* Willing to discontinue concomitant medications for CTCL for the duration of their study participation, including: high dose topical steroids - 2 week washout; oral steroids above 10 mg - 3 week washout; Psoralen + Ultraviolet A light (PUVA) or ultraviolet B light (UVB) (including sunbathing, tanning beds, etc.) - 2 week washout; extracorporeal photopheresis - 2 week washout; Electron Beam - 2 weeks washout; chemotherapeutic agents - 3 week washout; bexarotene capsules or other oral biologics - 2 week washout; and topical nitrogen mustard - 2 week washout.
* May re-enroll in the study if greater than 4 weeks elapses between courses and if all other inclusion/exclusion criteria are met.

Exclusion Criteria:

* Uncontrolled pain.
* Known history of autoimmune disease; or active HIV, HTLV-1, and/or hepatitis infection.
* Pregnant or lactating.
* Have sensitivity to drugs that provide local anesthesia.
* Have active malignancies with the exception of non-metastatic prostate cancer and carcinoma in situ of the skin and cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the micro array needle doxorubicin (MNA-D) system confirmed by vital signs, hematology, comprehensive metabolic panel, assessment for skin toxicity, and adverse event evaluation. | 9 weeks
  A traditional 3 + 3 dose escalation design will be used in 4 dosage cohorts (25 ug, 50 ug, 100 ug, and 200 ug).

SECONDARY OUTCOMES:
Evaluate the clinical responses (i.e., effectiveness) by the MNA-D | 12 months
  We will evaluate local, locoregional, and distant tumor regression; characterize and compare treated skin and the tumor microenvironment before, during, and after therapy

OTHER OUTCOMES:
Evaluate the tumor immunity induced by the MNA-D | 12 months
  Generalized skin changes, tissue and blood will be analyzed for immunologic response to the MNA-D in treated and control control cutaneous T-cell lymphoma lesions

CONTACTS AND LOCATIONS:
Overall Officials: Oleg E Akilov, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Department of Dermatology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bediz B, Korkmaz E, Khilwani R, Donahue C, Erdos G, Falo LD Jr, Ozdoganlar OB. Dissolvable microneedle arrays for intradermal delivery of biologics: fabrication and application. Pharm Res. 2014 Jan;31(1):117-35. doi: 10.1007/s11095-013-1137-x. Epub 2013 Aug 1. PMID 23904139